CLINICAL TRIAL: NCT06384118
Title: Construction and Preliminary Verification of interventionImpact of an IMB Theory-based Health Education Intervention on Hypoglycemic Coping in Patients With Type 2 Diabetes: a Pilot Study
Brief Title: Effects of a Health Intervention on Hypoglycemic Coping : a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yating Liu (Other)
Responsible Party: Sponsor-Investigator, Yating Liu, supervisor nurse, Yangzhou University
Organization: Yangzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: YZUHL20220047
Record Dates: First submitted 2024-01-17; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes Mellitus; Hypoglycemia; Health Education
Keywords: type 2 diabetes mellitus; hypoglycemic; coping style; IMB theory
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia; Health Education

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Based on IMB Theory of Health Education A hypoglycemia coping intervention program based on IMB theory was implemented on top of the control group.
  Interventions: Behavioral: Impact of an IMB theory-based health education intervention on hypoglycemic coping in patients with type 2 diabetes: a pilot study
- the control group (No Intervention): General diabetes health education Patients were provided with regular medication guidance, dietary guidance, exercise guidance and popularization of related diabetes knowledge; regular daily blood glucose testing and recording; and timely answers to patients' clinical problems and psychological support.

INTERVENTIONS:
Behavioral: Impact of an IMB theory-based health education intervention on hypoglycemic coping in patients with type 2 diabetes: a pilot study — Based on IMB health education theory Questionnaire collection, face-to-face interview, and manual interpretation on the first day of admission; questionnaire collection, face-to-face interview, and manual interpretation on the first day of admission; hypoglycemia knowledge promotion on the second day; Peer experience sharing on the third day; access to WeChat group and knowledge pushing on the fourth day; hypoglycemia-related lectures and practical teaching on the fifth day, face-to-face teaching and development of blood glucose management plan. Hypoglycemia knowledge contest on the day before discharge; One week, two weeks and three weeks after discharge for WeChat push or phone call; WeChat push, phone call and questionnaire.
  Arms: intervention group

SUMMARY:
From August 2023 to January 2024, 100 patients with type 2 diabetes who met the inclusion and exclusion criteria were selected from the endocrinology department of The purpose of this study was to construct a hypoglycemia coping intervention program for type 2 diabetic patients based on the IMB theory and to investigate the feasibility, acceptability, and initial effects of the program.

DETAILED DESCRIPTION:
In this study, eligible participants were randomized in a 1:1 ratio into an intervention group (health education based on IMB theory given on top of regular diabetes health education) and a control group (regular diabetes health education), with a 4-week intervention period and a 8-week follow-up period, for a total of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the 2018 ADA medical standards for Diabetes diagnosis and treatment, are diagnosed with T2DM and use insulin or sulfonylurea drugs;
* Duration of diabetes mellitus ≥1 year
* Age ≥18 years old;
* A history of hypoglycemia in the past 6 months;
* Type 2 diabetes patients with hypoglycemia coping style questionnaire inclination, avoidance, compromise;
* Good communication and language skills;
* Have a smartphone and can use it;
* Voluntary participation in this study.

Exclusion Criteria:

* Patients with type 1 diabetes;
* Patients with type 2 diabetes combined with serious complications;
* Patients who have recently or are participating in other similar studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
The hypoglycemic coping style | Baseline, 4 weeks, 8 weeks and 12 weeks post-intervention
  The scale consists of 16 entries in 3 dimensions, which in this study are confrontation (entries 1, 6, 8, 11, 12, 15), avoidance (entries 2, 5, 7, 10, 13, 16), and submission (entries 3, 4, 9, 14), and each of the entries is rated on a Likert's 5 scale ranging from 0-4, with higher scores on the dimensions indicating a greater tendency toward this type of coping, and the scale's total Cronbach's alpha coefficient was 0.821.

SECONDARY OUTCOMES:
hypoglycemic fear behavioral | Baseline, 4 weeks, 8 weeks and 12 weeks post-intervention
  Hypoglycemia fear-behavior scale (HFS-BS) consists of 19 entries and is scored on a 5-point Likert scale from 1 to 5, with total scores ranging from 15 to 95, with the higher scores indicating that the patients' hypoglycemia fear-behavior is more pronounced, and the higher the level of fear of hypoglycemia. The higher the score, the more obvious the change in the patient's hypoglycemic fear behavior and the higher the degree of hypoglycemic fear.
Hypoglycemia fear worry | Baseline, 4 weeks, 8 weeks and 12 weeks post-intervention
  Hypoglycemia fear survey-worry scale (HFS-WS) was used to assess the patients' feelings about hypoglycemia in the past six months. The scale has 13 entries, and adopts Likert's 5-point scale, with scores ranging from 0-4 from the lowest to the highest, and the total score ranging from 0 to 52, with the higher the score, the more fearful the patients are about hypoglycemia.
Level of health information access behavior | Baseline, 4 weeks, 8 weeks and 12 weeks post-intervention
  The Cronbach's alpha coefficient of the scale was 0.866, and a Likert 5-point scale was used, and a standardized score of the scale score (Index Score=(actual total score/possible highest score)*100%) of greater than 50% was considered moderately high. Higher scores represent higher levels of health information acquisition behavior.
Level of health beliefs | Baseline, 4 weeks, 8 weeks and 12 weeks post-intervention
  The questionnaire consisted of 20 items in 5 latitudes, mainly for the necessity of diabetes treatment, benefits, harms, hazards of diabetes, and motivation to maintain the health of the organism, and the Cronbach's alpha coefficient of the scale was 0.89, and the questionnaire was scored on a 5-point Likert scale, with 8 to 14 being inverse scores, and the higher the total score indicated that the patient's beliefs about health were stronger.
Level of diabetes knowledge | Baseline, 4 weeks, 8 weeks and 12 weeks post-intervention
  The Cronbach's alpha coefficient of the questionnaire was 0.909, and the factor rotation analysis extracted six main factors explaining basic knowledge , dietary knowledge, exercise knowledge, self-monitoring knowledge, medication knowledge and complication knowledge. The variance explained by individual factors was above 7%, and the cumulative variance contribution rate was 69.004%, indicating that the questionnaire had good internal consistency. The evaluation standard of the questionnaire was 1 point for a correct answer, 0 point for an incorrect or unclear answer, and the cumulative score of the 34 items was added to the total knowledge score, and the higher the score, the more knowledge about diabetes mellitus was acquired.

CONTACTS AND LOCATIONS:
Overall Officials: Ya T Liu, Bachelor, Principal Investigator — Yangzhou University
Locations (1):
- Ya ting Liu, Yangzhou, 未选择, China

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT06384118/Prot_SAP_000.pdf